CLINICAL TRIAL: NCT05519579
Title: Intrathecal Chemoprophylaxis to Prevent Neurotoxicity Associated With Blinatumomab Therapy for Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NSH 1354
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Methotrexate; blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intrathecal chemotherapy before blinatumomab (Experimental)
  Interventions: Drug: Methotrexate; Drug: Blinatumomab

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 12mg given intrathecally within 24 hours prior to blinatumomab administration
Drug: Blinatumomab — Blinatumomab 28ug/day continuous infusion for 4 weeks

SUMMARY:
Changing the schedule of intrathecal chemotherapy to be given before and during blinatumomab will maintain the anti-leukemic effects of this drug while at the same time adding the benefit of limiting the neurotoxicity associated with cytokine release.

ELIGIBILITY:
Inclusion Criteria:

* Adults receiving first cycle of blinatumomab for relapse/refractory or MRD-positive B-cell Acute Lymphoblastic Leukemia
* Adequate renal and hepatic function
* Negative for HIV
* Negative serum pregnancy test, if applicable
* ECOG 0-2

Exclusion Criteria:

* Active CNS involvement by ALL
* Relative CNS disorders (seizure, paresis, aphasia, Cerebrovascular ischemia/hemorrhage, severe brain injury, dementia, Parkinson's, cerebellar disease, psychosis, coordination or movement disorder)
* Contraindication to receive intrathecal methotrexate
* Prior treatment with blinatumomab
* Active malignancy other than ALL
* Active infection or any other concurrent disease or medical condition that was deemed to interfere with the conduct of the study as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that experienced neurotoxicity during the first cycle of blinatumomab therapy | 28 days after first infusion
  Record occurrence and severity of neurotoxicity based on CTCAE criteria

SECONDARY OUTCOMES:
Number of participants that experienced cytokine release syndrome during the first cycle of blinatumomab therapy | 28 days after first infusion
  Record occurrence and severity of cytokine release syndrome based on CTCAE criteria
Number of participants with a response of complete remission and MRD negativity at the end of cycle 1 | 28 days after first infusion
  Conduct disease restaging assessments, such as bone marrow biopsies and lumbar punctures, to determine response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Melhem Solh, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kantarjian H, Stein A, Gokbuget N, Fielding AK, Schuh AC, Ribera JM, Wei A, Dombret H, Foa R, Bassan R, Arslan O, Sanz MA, Bergeron J, Demirkan F, Lech-Maranda E, Rambaldi A, Thomas X, Horst HA, Bruggemann M, Klapper W, Wood BL, Fleishman A, Nagorsen D, Holland C, Zimmerman Z, Topp MS. Blinatumomab versus Chemotherapy for Advanced Acute Lymphoblastic Leukemia. N Engl J Med. 2017 Mar 2;376(9):836-847. doi: 10.1056/NEJMoa1609783. PMID 28249141
- [Background] Gokbuget N, Dombret H, Bonifacio M, Reichle A, Graux C, Faul C, Diedrich H, Topp MS, Bruggemann M, Horst HA, Havelange V, Stieglmaier J, Wessels H, Haddad V, Benjamin JE, Zugmaier G, Nagorsen D, Bargou RC. Blinatumomab for minimal residual disease in adults with B-cell precursor acute lymphoblastic leukemia. Blood. 2018 Apr 5;131(14):1522-1531. doi: 10.1182/blood-2017-08-798322. Epub 2018 Jan 22. PMID 29358182
- [Background] Topp MS, Gokbuget N, Zugmaier G, Klappers P, Stelljes M, Neumann S, Viardot A, Marks R, Diedrich H, Faul C, Reichle A, Horst HA, Bruggemann M, Wessiepe D, Holland C, Alekar S, Mergen N, Einsele H, Hoelzer D, Bargou RC. Phase II trial of the anti-CD19 bispecific T cell-engager blinatumomab shows hematologic and molecular remissions in patients with relapsed or refractory B-precursor acute lymphoblastic leukemia. J Clin Oncol. 2014 Dec 20;32(36):4134-40. doi: 10.1200/JCO.2014.56.3247. Epub 2014 Nov 10. PMID 25385737
- [Background] Topp MS, Gokbuget N, Stein AS, Zugmaier G, O'Brien S, Bargou RC, Dombret H, Fielding AK, Heffner L, Larson RA, Neumann S, Foa R, Litzow M, Ribera JM, Rambaldi A, Schiller G, Bruggemann M, Horst HA, Holland C, Jia C, Maniar T, Huber B, Nagorsen D, Forman SJ, Kantarjian HM. Safety and activity of blinatumomab for adult patients with relapsed or refractory B-precursor acute lymphoblastic leukaemia: a multicentre, single-arm, phase 2 study. Lancet Oncol. 2015 Jan;16(1):57-66. doi: 10.1016/S1470-2045(14)71170-2. Epub 2014 Dec 16. PMID 25524800
- [Background] Bargou R, Leo E, Zugmaier G, Klinger M, Goebeler M, Knop S, Noppeney R, Viardot A, Hess G, Schuler M, Einsele H, Brandl C, Wolf A, Kirchinger P, Klappers P, Schmidt M, Riethmuller G, Reinhardt C, Baeuerle PA, Kufer P. Tumor regression in cancer patients by very low doses of a T cell-engaging antibody. Science. 2008 Aug 15;321(5891):974-7. doi: 10.1126/science.1158545. PMID 18703743
- [Background] Topp MS, Kufer P, Gokbuget N, Goebeler M, Klinger M, Neumann S, Horst HA, Raff T, Viardot A, Schmid M, Stelljes M, Schaich M, Degenhard E, Kohne-Volland R, Bruggemann M, Ottmann O, Pfeifer H, Burmeister T, Nagorsen D, Schmidt M, Lutterbuese R, Reinhardt C, Baeuerle PA, Kneba M, Einsele H, Riethmuller G, Hoelzer D, Zugmaier G, Bargou RC. Targeted therapy with the T-cell-engaging antibody blinatumomab of chemotherapy-refractory minimal residual disease in B-lineage acute lymphoblastic leukemia patients results in high response rate and prolonged leukemia-free survival. J Clin Oncol. 2011 Jun 20;29(18):2493-8. doi: 10.1200/JCO.2010.32.7270. Epub 2011 May 16. PMID 21576633
- [Background] Martinelli G, Boissel N, Chevallier P, Ottmann O, Gokbuget N, Topp MS, Fielding AK, Rambaldi A, Ritchie EK, Papayannidis C, Sterling LR, Benjamin J, Stein A. Complete Hematologic and Molecular Response in Adult Patients With Relapsed/Refractory Philadelphia Chromosome-Positive B-Precursor Acute Lymphoblastic Leukemia Following Treatment With Blinatumomab: Results From a Phase II, Single-Arm, Multicenter Study. J Clin Oncol. 2017 Jun 1;35(16):1795-1802. doi: 10.1200/JCO.2016.69.3531. Epub 2017 Mar 29. PMID 28355115
- [Background] Jain T, Litzow MR. No free rides: management of toxicities of novel immunotherapies in ALL, including financial. Blood Adv. 2018 Nov 27;2(22):3393-3403. doi: 10.1182/bloodadvances.2018020198. PMID 30482769
- [Background] Shah NN, Johnson BD, Fenske TS, Raj RV, Hari P. Intrathecal chemotherapy for management of steroid-refractory CAR T-cell-associated neurotoxicity syndrome. Blood Adv. 2020 May 26;4(10):2119-2122. doi: 10.1182/bloodadvances.2020001626. No abstract available. PMID 32407473